CLINICAL TRIAL: NCT00035880
Title: A Phase II/III, Multicenter, Open Label, Randomized Clinical Trial Evaluating ABX-CBL When Compared to Atgam as Second Line Therapy in Patients With Steroid Resistant Acute Graft Versus Host Disease
Brief Title: Study Comparing ABX-CBL (Monoclonal Antibody) Versus Atgam in Patients With Steroid Resistant Acute Graft Versus Host Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abgenix (Industry)
Collaborators: Sangstat Medical Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABX-CB-9906; NCT00012077 (obsolete NCT alias)
Record Dates: First submitted 2002-05-06; First posted 2002-05-07 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-07

CONDITIONS: Graft Vs Host Disease
Keywords: Acute graft versus host disease; Stem Cell Transplantation
MeSH Terms: conditions — Graft vs Host Disease

INTERVENTIONS:
Drug: ABX-CBL

SUMMARY:
Trial evaluating the improvement in survival at 180 days of two therapies (Atgam versus ABX-CBL, a monoclonal antibody) in patients with acute graft versus host disease that does not respond to steroid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of single allogeneic stem cell transplant from any donor type
* Time post transplant less than 100 days
* Received no treatment for GVHD other than steroids

Exclusion Criteria:

* Recipient of second allogeneic stem cell transplant or subsequent lymphocyte product from the donor post transplant
* IBMTR index less than A
* Received any murine product in the past
* Diagnosed with chronic GVHD
* Received Atgam later than day 10 post transplant
* Change to prophylactic regimen for acute GVHD within 72 hours of randomization

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95
Dates: Start 1999-10; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Locations (1):
- Abgenix, Inc, Fremont, California, United States